CLINICAL TRIAL: NCT04298502
Title: The Molecular Mechanism of CMV-driven NKG2C+NK Cell Expansion in Human
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Head of Peking University Institute of Hematology, Peking University People's Hospital
Other Study IDs: HCMV-NKG2C+ NK cell
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Acute Leukemia; CMV Viremia; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observation study to investigate the molecular mechanism of NKG2C+NK cell expansion after HCMV infection

DETAILED DESCRIPTION:
According to the changes of molecular and gene expression in NK cells at different time points after infection, we want to find out the mechanism by which HCMV promotes the expansion of NKG2C + NK cells.

ELIGIBILITY:
Inclusion Criteria:

1. AML or MDS or CML or ALL undergoing haploidentical stem cells transplantation
2. No severe organ dysfunction or failure
3. Subjects must be capable of, and willing to provide written informed consent to participate in the study. Subjects unable to provide written informed consent by themselves may be consented through their legal representative.

Exclusion Criteria:

1. Participation in another industry-sponsored clinical study where treatment for CMV is already specified by the study protocol.
2. Patients received other adoptive immunotherapy such as donor lymphocyte infusion (DLI), Epstein-Barr virus (EBV)-specific T cells and so on.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AML or MDS or CML or ALL undergoing haploidentical stem cells transplantation AND the healthy donors.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
CMV viremia | 2 moths post-transplantation
  CMV-DNA>1.0x10^3 cpies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, M.D., PhD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China